CLINICAL TRIAL: NCT04987593
Title: Characterisation of the Gut Microbiota in Term Infants After Maternal Prenatal and Postnatal Supplementation of Probiotics - an Open Label Pilot Study
Brief Title: Characterisation of the Gut Microbiota in Term Infants After Maternal Supplementation of Probiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chr Hansen (Industry)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Organization: ChrHansen (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HND-IN-039
Record Dates: First submitted 2021-06-29; First posted 2021-08-03 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2021-08

CONDITIONS: Infant Development; Gut Microbiome
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Four probiotic strains to be consumed once daily
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — Once a day daily intake of probiotics, at least for 28 consecutive days before giving birth and for at least 28 consecutive days after giving birth

SUMMARY:
A monocenter, open label pilot study in pregnant women and their offspring with at least four weeks prenatal and four weeks postnatal maternal intervention with a study product consisting of four different food constituents.

The study will investigate the effect of maternal supplementation with the food constituents on the recovery of the constituents in the maternal and infant feces, the microbiota in both mother and infant and potential transmission routes from mother to infant.

DETAILED DESCRIPTION:
Pregnant women will be recruited at the ordinary midwife visit in gestational week 28. The intervention will begin in gestational week 33+0 to ensure at least four weeks prenatal intervention before expected birth.

The study will be conducted in four phases. First phase is the run-in phase. The second phase is the prenatal intervention period from gestational week 33+0 until birth. Third phase is the postnatal intervention period, from birth until four weeks postnatal. The last phase is a two weeks follow-up period without any intake of the investigational product.

Infant stool samples, as well as maternal breast milk samples, stool and urine samples and samples from vagina will be collected on multiple occasions during the study. In addition, sample from placenta, umbilical cord, umbilical cord blood and amnion fluid will be collected. Mothers will be asked to complete electronic questionnaires daily during the course of the study.

ELIGIBILITY:
Inclusion Criteria

Pregnant women:

1. Enrolled at Aarhus University Hospital
2. Singleton pregnancy
3. Age above 18 years at informed consent
4. Aim to give birth vaginally
5. Aim to breastfeed
6. No use of probiotics (contained in dietary supplements/ food) after written consent.

Infants:

1. Gestational age between 37-42 weeks

Exclusion Criteria:

Pregnant women • Use of immunosuppressant drugs.

Infants:

• None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Recovery of study product in infant feces | 28 days after birth
  Presence of at least one of the probiotic strains in infant feces using PCR

SECONDARY OUTCOMES:
Recovery of study product in maternal feces | 28 days
  Presence of at least one of the probiotic strains in maternal feces using PCR
Quantification of the microbiota in breastmilk | 28 days after birth
  Characterization of breastmilk microbiota by and recovery of probiotic strains using PCR
Quantification of the maternal vaginal microbiota | 28 days
  Characterization of the vaginal microbiota and recovery of probiotic strains using PCR

OTHER OUTCOMES:
Infant gastrointestinal problems | 28 days
  Infants gastrointestinal problems will be assessed using the Parent-Report Form for Neonates Section A - Infant Gastrointestinal Problems (ROME IV)
Infant stool frequency and consistency | 28 days
  Infants stool frequency and consistency will be assessed using Amsterdam Stool Chart
Infant Reflux | 28 days
  Reflux will be assessed using the Infant Gastroesophageal Reflux Questionnaire Revised (I-GERQ-R)
Adverse events | 12 weeks
  Any adverse events experienced by either mother or infant will be recorded during the entire study period

CONTACTS AND LOCATIONS:
Overall Officials: Lars Henning Pedersen, MD, Principal Investigator — Department of Gynecology and Obstetrics, Aarhus University Hospital
Locations (1):
- Department of Gynaecology and Obstetrics, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
No IPD plan yet